CLINICAL TRIAL: NCT06263595
Title: Mitigating Harm: Assessing Preoperative Residual Gastric Volumes to Risk Stratify Patients Administering Semaglutide
Brief Title: Semaglutide and Preoperative Residual Gastric Volumes
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Joanna Moser, Clinical Assistant Professor, University of Calgary
Other Study IDs: REB23-1754
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLP-1 Agonist Group: Intervention: elective surgical patients taking GLP-1 receptor agonists
  Interventions: Device: gastric antral sonography
- Non GLP-1 Agonist Group: Intervention: elective surgical patients not taking GLP-1 receptor agonists
  Interventions: Device: gastric antral sonography

INTERVENTIONS:
Device: gastric antral sonography — Participant will undergo gastric antrum ultrasound and be scanned in the supine position followed by the right lateral decubitus position. Qualitative and quantitative assessments will be completed.

SUMMARY:
Given the pharmacodynamic and pharmacokinetic properties of glucagon-like peptide-1 (GLP-1) agonists, the Canadian Anesthesiologists' Society has recognized that patients on GLP-1 agonists may have an increased aspiration risk due to a 'full stomach,' even after following preoperative fasting guidelines. In other words, safe fasting timelines are not known in individuals taking GLP-1 agonists, as demonstrated by recent case reports of patients who either retained or regurgitated stomach contents despite being adequately fasted.

To address this gap, we plan to measure preoperative residual gastric volumes with point-of-care ultrasound (POCUS) in patients taking this medication. The priority is to first gather data to identify which patient populations need risk stratification and to then use this data to support the development of specific guidelines that reduce anesthetic complications, such as aspiration pneumonia.

Our primary objective is to use POCUS preoperatively to assess gastric volumes of fasted patients to demonstrate if there is a clinically significant increase in residual gastric volumes in patients on semaglutide.

ELIGIBILITY:
Inclusion Criteria:

* all elective surgical patients (> 18 years of age)
* followed institutional fasting protocol for surgery
* patients taking GLP-1 receptor agonist (subcutaneous for weight management and/or blood glucose control in type II diabetes mellitus, N = 45)
* patients not taking GLP-1 receptor agonist (N =45)

Exclusion Criteria:

* confounding delayed gastric emptying due to pregnancy
* previous esophageal or gastric operation
* etiologies at increased risk for delayed gastric emptying (hiatal hernia, Parkinson's disease, scleroderma, multiple sclerosis, and amyloidosis)
* on medication that could potentially cause gastroparesis or delayed gastric or intestinal emptying (opioids, proton pump inhibitors, tricyclic antidepressants, calcium channel blockers, antipsychotic medications, loperamide, diphenoxylate, oxybutynin, hyoscine butylbromide, scopolamine, promethazine, glycopyrrolate, atropine, chlordiazepoxide, and lithium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients meeting inclusion/exclusion criteria at the South Health Campus (Calgary, AB, Canada)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants presenting with a full stomach | Measured in the preoperative holding area
  Full stomach defined as either clear fluid > 1.5ml/kg or solid content found with point-of-care gastric antral sonography.

SECONDARY OUTCOMES:
Number of occurrences requiring change in anesthetic management plan | From time of preoperative ultrasound in holding area to anesthesia induction in operating room
  Changes in plan include those from laryngeal mask airway to more advanced endotracheal tube with rapid sequence induction and intubation or spinal anesthetic without sedation to administration of a general anesthetic.
Relationship between dose, duration and timing of GLP-1 receptor agonist and gastric volume | Measured in the preoperative holding area
  Explore if dose, duration, and timing of GLP-1 receptor agonist affects gastric volume
Relationship between gastric emptying and purpose of GLP-1 receptor agonist administration | Measured in the preoperative holding area
  Explore if GLP-1 receptor agonist impacts gastric emptying different in patients administering for Type II diabetes mellitus or weight management

CONTACTS AND LOCATIONS:
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No